CLINICAL TRIAL: NCT05940025
Title: Multidisciplinary Digital Therapeutics for Chronic Low Back Pain Versus In-person Education Combined With Physiotherapy, a Randomized Controlled Pilot Study
Brief Title: Multidisciplinary Digital Therapeutics of Chronic Lower Back Pain Versus Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EverEx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-ETH-02K-CTP-01
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MORT-LBP (Experimental): Participants randomly assigned to this arm will use the app, MORT-LBP.
  Interventions: Device: MORT-LBP
- treatment as usual (TAU) (Active Comparator): Participants randomly assigned to this arm will receive their TAU only (no use of the app, MORT-LBP).
  Interventions: Other: treatment as usual (TAU)

INTERVENTIONS:
Device: MORT-LBP — The MORT-LBP, developed by EverEx, Inc., is designed to provide multidisciplinary rehabilitation treatment, a combination of graded exercise therapy and cognitive behavioral therapy for patients with chronic lower back pain.
  Arms: MORT-LBP
Other: treatment as usual (TAU) — In the control group, education and physiotherapy is delivered and self-exercise is recommended.
  Arms: treatment as usual (TAU)

SUMMARY:
This randomized controlled pilot study will be evaluating an app, MORT-LBP app (ETH-02K), owned by EverEx, Inc., to examine safety and efficacy in individuals with chronic lower back pain.

DETAILED DESCRIPTION:
This randomized controlled pilot study will enroll 46 participants, where half will be randomly assigned to the app, MORT-LBP (n = 23), and half will be assigned to treatment as usual (TAU) (n = 23), to examine safety and efficacy in individuals with chronic lower back pain. All subjects will be followed up in the study for a total of 12 weeks, 8-week courses of treatment with additional 4-week observation. The app provides multidisciplinary rehabilitation treatment, a combination of graded exercise therapy and cognitive behavioural therapy for patients with chronic lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 19 and <65 years of age
* Patients who have a history of lower back pain persisting for longer than 12 weeks
* Patients who have average back pain score of 3 or more on the numeric rating scale (NRS)
* Patients who can use application-based therapy with his/her smartphone
* Patients who signed a written informed consent form
* Patients who are able to comply with the plan, as determined by the study investigator.

Exclusion Criteria:

* Patients who have previous history of spinal surgery
* Patients who have previous history of spinal trauma within 3 months
* Patients with lower extremity radicular pain with sensory and motor dysfunction
* Patients with lower extremity muscle strength of 3 or less on a manual muscle test
* Patients with spondylolysis or spondylolisthesis
* Patients with other structural abnormalities of the spine, including scoliosis (Cobb's angle > 10 degrees) or kyphosis (lordotic angle < 0 degrees)
* Patients with red flag signs (paralyzing symptoms such as fecal impairment, sudden unexplained weight loss)
* Patients with tumors, infections, metabolic bone disease, cognitive impairment, fibromyalgia, and systemic inflammatory diseases
* Patients with other systemic disease conditions that limit exercise therapy, as determined by the study investigator
* Patients who are pregnant or breastfeeding
* Patients with known substance/alcohol use disorders
* Patients who are not able to participate in an exercise or strengthening program
* Patients taking opioid analgesic medications with a potency greater than or equal to tramadol for other conditions or low back pain

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Usual pain severity in the past week assessed by the Numeric Rating Scale (NRS) | 8 weeks
  The primary outcome being measure is differences in usual pain severity in the past week between groups after the intervention. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Worst pain severity in the past week assessed by the Numeric Rating Scale (NRS) | 8 weeks
  The primary outcome being measure is differences in worst pain severity in the past week between groups after the intervention. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Functional disability assessed by Oswestry Disability Index (ODI) | 8 weeks
  The primary outcome being measure is differences in functional disability between groups after the intervention. Oswestry Disability Index (ODI) is a patient reported assessment of chronic lower back pain-specific functional limitations. It has 10 questions, total score ranging from 0 to 50, and ODI is calculated with (total score)/(answered question number * 5)*100%. Higher index means worse outcome.

SECONDARY OUTCOMES:
Ususal pain severity in the past week assessed by Numeric Rating Scale (NRS) | 4, 12 weeks
  The secondary outcome being measure is differences in usual pain severity in the past week between groups at 4 and 12 weeks. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Worst pain severity in the past week assessed by Numeric Rating Scale (NRS) | 4, 12 weeks
  The secondary outcome being measure is differences in worst pain severity in the past week between groups at 4 and 12 weeks. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Functional disability assessed by Oswestry Disability Index (ODI) | 4, 12 weeks
  The secondary outcome being measure is differences in functional disability between groups at 4 and 12 weeks. Oswestry Disability Index (ODI) is a patient reported assessment of chronic lower back pain-specific functional limitations. It has 10 questions, total score ranging from 0 to 50, and ODI is calculated with (total score)/(answered question number * 5)*100%. Higher index means worse outcome.
Health-related quality of life assessed by EuroQol five-dimensional (EQ-5D) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in health-related quality of life between groups at 4, 8 and 12 weeks. It measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with three possible answers for each dimension (1=no problem, 2=moderate problem, 3=severe problem). The instrument also includes a visual analogue scale, which is numbered from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Assessment of mental health symptoms specific to depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 8, 12 weeks
  Differences in mental health symptoms between groups at 8, 12 weeks. The Patient Health Questionnaire-9 (PHQ-9) total score for the nine items ranges from 0 to 27 (higher scores indicating greater severity of depression).
Assessment of catastrophic thinking measured by Pain Catastrophizing Scale (PCS) | 8, 12 weeks
  Differences in levels of catastrophic thinking between groups at 8, 12 weeks. The Pain Catastrophizing Scale (PCS) is a 13-item scale, with a total range of 0 to 52 (higher scores indicating higher amounts of pain catastrophizing).
Assessment of fear avoidance behaviours measured by Fear-Avoidance Beliefs Questionnaire (FABQ) | 8, 12 weeks
  Differences in fear avoidance behaviours between groups at 8, 12 weeks. The Fear-Avoidance Beliefs Questionnaire (FABQ) is a 16-item scale, with a total range of 0 to 96 (higher scores indicating higher amounts of fear avoidance behaviours).
Assessment of spinal alignment status measured by X-ray | 8 weeks
  Differences in Cobb's angle, distances from the plumb line of C7, lumbar lordosis, pelvic tilt, pelvic incidence, sacral slope, and distances from the plumb line of C7 and posterosuperior edge of S1 vertebral body between group after intervention.
Assessment of Equilibrium Ability by Single-limb stance test | 4, 8, 12 weeks
  Differences in single-limb stance test between group at 4, 8, 12 weeks. The single limb stance test measures how long a individual can stand on each leg for up to 20 seconds.
Assessment of Muscular Endurance by Prone bridge test and Borg CR10 Scale (2010) | 4, 8, 12 weeks
  Differences in prone bridge test test between group at 4, 8, 12 weeks. The prone bridge test measures how long a individual can stand prone bridge test for up to 120 seconds. Afterward, Borg CR10 Scale (2010), the rating of perceived exertion after physical activity is measured. It ranges from 0 to 10 (higher scores indicating more sensation of hardness).
Changes of usual and worst pain severity in the past week assessed by Numeric Rating Scale (NRS) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in changes of usual pain severity, worst pain severity, Oswestry Disability Index (ODI), EuroQol five-dimensional (EQ-5D), Single-limb stance test, Prone bridge test and Borg CR10 Scale (2010) from baseline to 4, 8, and 12 weeks between groups. NRS score was measured from 0 (no pain) to 10 (worst pain imaginable).
Changes of Oswestry Disability Index (ODI) and EuroQol five-dimensional (EQ-5D) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in changes of Oswestry Disability Index (ODI) and EuroQol five-dimensional (EQ-5D) from baseline to 4, 8, and 12 weeks between groups. Oswestry Disability Index (ODI) is a patient reported assessment of chronic lower back pain-specific functional limitations. It has 10 questions, total score ranging from 0 to 50, and ODI is calculated with (total score)/(answered question number * 5)*100%. Higher index means worse outcome. EQ-5D measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with three possible answers for each dimension (1=no problem, 2=moderate problem, 3=severe problem). The instrument also includes a visual analogue scale, which is numbered from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Changes of Single-limb stance test, Prone bridge test and Borg CR10 Scale (2010) | 4, 8, 12 weeks
  The secondary outcome being measure is differences in changes of single-limb stance test, prone bridge test and Borg CR10 Scale (2010) from baseline to 4, 8, and 12 weeks between groups. The single limb stance test measures how long a individual can stand on each leg for up to 20 seconds. The prone bridge test measures how long a individual can stand prone bridge test for up to 120 seconds. Afterward, Borg CR10 Scale (2010), the rating of perceived exertion after physical activity is measured. It ranges from 0 to 10 (higher scores indicating more sensation of hardness).
Use of rescue medication | 4, 8, 12 weeks
  Differences in use of rescue medication between groups at 4, 8, 12 weeks.
Assessment of retention in treatment | 4, 8 weeks
  Differences in retention rates between groups at 4, 8 weeks.
Assessment of app usability by surveys | 4, 8 weeks
  Differences in app usability survey score between groups at 4, 8 weeks. The survey comprises 8 questions, with total score ranging from 0 to 40. Higher score indicates better user experience.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Yeol Chang, M.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Hanyang University Guri Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No